CLINICAL TRIAL: NCT01939912
Title: Study on Reflex Response During Temporary Stimulation and Inhibition of Chemoreceptors of Carotid Bodies - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noblewell (Industry)
Collaborators: Cibiem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADENOSINE-PILOT-CIBIEM
Record Dates: First submitted 2013-08-29; First posted 2013-09-11 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure; Peripheral Chemoreceptor Hypersensitivity
MeSH Terms: conditions — Heart Failure | interventions — Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stimulation of carotid body chemoreceptors (Experimental): Adenosine boluses will be administered through an intravascular catheter used to administer the contrast agent during the carotid artery arteriography.
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — Antiarrhythmic agent.

SUMMARY:
The isolated response of the carotid bodies to local stimulation with adenosine has not been researched in humans. There are single reports indicating that intravenous administration of adenosine causes hyperventilation through activating the carotid bodies.

Adenosine will be injected intraarterially during invasive treatment (percutaneous carotid artery stenting, CAS) or diagnostic (arteriography) procedures and their conduct will only slightly influence the standard scheme of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* stenosis of one of the internal carotid arteries qualifying the patient to the procedure treatment (according to the ESC 2011 or American Heart Association (AHA) guidelines) or the necessity of the carotid artery arteriography, in order to verify the level of narrowing;
* in the case of procedure treatment, patient's declaration to be treated by the percutaneous method;
* stable clinical condition for at least 4 weeks prior to the inclusion in the study;
* over 18 years of age;
* ability to give and giving the informed consent to participate in the study.

Exclusion Criteria:

* bilateral significant carotid artery stenosis;
* complete closure or critical constriction of either of the carotid arteries;
* brain stroke or transient ischaemic attack (TIA) within 6 months prior to the inclusion in the study;
* unstable angina pectoris, coronary attack within 3 months prior to the inclusion in the study;
* coronary revascularisation or clinically significant infection within 1 month prior to the inclusion in the study;
* significant chronic neurological condition in medical history;
* dipyridamole or theophyline-based medications taken by the patient;
* bronchial asthma;
* GOLD 3 or 4 Chronic Obstructive Pulmonary Disease (COPD) in medical history;
* second or third degree atrioventricular block, sick sinus syndrome, or an additional evident track of atrioventricular conducting;
* advanced first degree atrioventricular block (PQ > 240 ms)
* extension of the QTc interval > 0.5 s;
* grade 3 (ESC) arterial hypertension;
* previously stated oversensitivity to adenosine;
* pregnancy;
* patients undergoing haemodialysis or peritoneal dialysis at inclusion in the study;
* undergone heart transplantation;
* any significant, in the investigator's assessment, aberrations detected in additional tests, increasing the risk related to performing procedures predicted by the protocol;
* lack of informed consent for the participation in the study;
* stage III (Fontaine) obliterative arteriosclerosis of the lower limb and/or Buerger's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Ventilation at rest | 30 minutes
  Assessment of the adenosine influence on the monitored parameter
Arterial blood pressure | 30 minutes
  Assessment of the adenosine influence on the monitored parameter

SECONDARY OUTCOMES:
ECG | 30 minutes
  Assessment of the adenosine influence on the monitored parameter
Capillary blood saturation | 30 minutes
  Assessment of the adenosine influence on the monitored parameter
Breathing pattern | 30 minutes
  Assessment of the adenosine influence on the monitored parameter

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Ponikowski, Prof., Principal Investigator — 4. Wojskowy Szpital Kliniczny we Wroclawiu
Locations (1):
- Centrum Chorób Serca - Klinika Kardiologii, 4. Wojskowy Szpital Kliniczny, Wroclaw, Poland

REFERENCES:
- [Derived] Tubek S, Niewinski P, Reczuch K, Janczak D, Rucinski A, Paleczny B, Engelman ZJ, Banasiak W, Paton JF, Ponikowski P. Effects of selective carotid body stimulation with adenosine in conscious humans. J Physiol. 2016 Nov 1;594(21):6225-6240. doi: 10.1113/JP272109. Epub 2016 Sep 11. PMID 27435894